CLINICAL TRIAL: NCT02473497
Title: CRIZOTINIB (XALKORI(REGISTERED)) EXPANDED ACCESS PROTOCOL FOR THE TREATMENT OF ADULT OR PEDIATRIC PATIENTS WITH SOLID OR HEMATOLOGIC MALIGNANCIES THAT HARBOR A CRIZOTINIB-SENSITIVE MOLECULAR ALTERATION BUT WHO ARE UNABLE TO SWALLOW CRIZOTINIB CAPSULES
Brief Title: Crizotinib (Xalkori) Expanded Access Protocol For The Treatment Of Adult Or Pediatric Patients
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A8081056; A8081056 (Other: Alias Study Number)
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Neoplasm
Keywords: chromosomal rearrangement; activating mutation; activating genetic alteration; genetic aberration; ALK; ROS1; cMET; crizotinib; oral formulation
MeSH Terms: conditions — Neoplasms | interventions — Crizotinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Crizotinib — For adult patients, crizotinib 250 mg BID will be administered orally at approximately the same time each day on a continuous daily dosing schedule, ie, without break in dosing. For pediatric patients, crizotinib 280 mg/m2 BID will be administered orally at approximately the same time each day on a continuous daily dosing schedule, ie, without break in dosing.
  Other Names: XALKORI

SUMMARY:
This is an open label expanded access protocol for the treatment of up to approximately 40 adult or pediatric (defined as age <18 years) patients with tumors harboring either a chromosomal translocation or activating mutation involving the ALK or ROS1 gene or an activating genetic alteration involving the cMET gene who cannot swallow the crizotinib capsule but may be able to derive benefit from treatment with an alternative oral formulation of crizotinib.

DETAILED DESCRIPTION:
Crizotinib is indicated in the U.S. for the treatment of patients with metastatic non-small cell lung cancer (NSCLC) whose tumors are anaplastic lymphoma kinase (ALK)-positive as detected by an FDA-approved test. Commercially available dosage forms are 250 mg and 200 mg capsules. This expanded access protocol (EAP) is designed to provide access to an alternative oral formulation of crizotinib for those patients who are unable to swallow capsules.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of a primary or metastatic malignancy that is positive for a chromosomal translocation or activating mutation involving the ALK or ROS1 gene or an activating genetic alteration involving the c MET gene, as determined by local clinical testing that is appropriately validated in accordance with applicable regulatory guidelines and/or practice standards (patients with tumors harbouring other genetic alterations that may potentially benefit from treatment with crizotinib eg NTRK3 ETV6 fusion gene may be considered on a case by case basis subject to approval by the sponsor).
* Inability to swallow crizotinib capsules, adult patients of whom must either have a feeding tube in place or have completed clinical evaluation of dysphagia without any reversible causes identified.
* At least 12 months of age (patients <12 months of age will be evaluated on a case by case basis and discussed with the sponsor).

Exclusion Criteria:

* Currently receiving crizotinib, another ALK inhibitor, or an investigational product.
* Adult patients who have been previously treated with crizotinib.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (16):
  - Children's Hospital Colorado, Aurora, Colorado
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - West Chester Medical Center, Hawthorne, New York
  - Cohen Children's Medical Center of New York, New Hyde Park, New York
  - New York Medical College, Valhalla, New York
  - Westchester Medical Center/Maria Fareri Children's Hospital, Valhalla, New York
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia (Investigational Pharmacy), Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A8081056